CLINICAL TRIAL: NCT03030066
Title: A Phase 1 Study of DS-1001b in Patients With IDH1 Mutated Gliomas
Brief Title: Study of DS-1001b in Patients With Gene IDH1-Mutated Gliomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS1001-A-J101; 163479 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glioma
Keywords: DS-1001b; IDH1 mutation; Developmental Phase I; Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Drug DS-1001b (Experimental): Oral administration
  Interventions: Drug: DS-1001b

INTERVENTIONS:
Drug: DS-1001b — Generic not assigned
  Other Names: Investigational

SUMMARY:
This is a study to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and anti-tumor activity of DS-1001b in patients with gliomas that harbor IDH1-R132 mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically confirmed glioma with an IDH1-R132 mutation
2. Has disease that has recurred or progressed following standard treatment including radiotherapy
3. Has measurable lesion(s) as per RANO criteria
4. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

Exclusion Criteria:

1. Has significant symptoms of increased intracranial pressure
2. Has another active neoplasm
3. Has active infection requiring systemic treatment
4. Has a history of severe cardiac disease
5. Has had prior treatment with any inhibitor targeting mutant IDH1
6. Has had investigational drug treatment within 4 weeks prior to the first dose of study treatment
7. Is a pregnant or lactating female

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with dose limiting toxicities | 21 days

SECONDARY OUTCOMES:
Percentage of participants experiencing an adverse event (AE) | up to 36 months
  AEs temporally associated with DS-1001b treatment
Area under the concentration curve (AUC) for DS-1001b | up to 36 months
Maximum plasma concentration (Cmax) for DS-1001b | up to 36 months
Time to maximum plasma concentration (Tmax) for DS-1001b | up to 36 months
Change from baseline in 2-hydroxyglutarate (2-HG) concentration in patient specimens after treatment with DS-1001b | Baseline, up to 36 months
Tumor response to DS-1001b based on Response Assessment in Neuro-Oncology Criteria (RANO) | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- National Cancer Center Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/